CLINICAL TRIAL: NCT02708485
Title: Evaluating the Impact of Physical Exercise on Mild Alzheimer's Disease in a Randomized Clinical Trial: Quantification With 18F -FDG and 11C- AcAc PET Imaging
Brief Title: Effect of Walking on Brain Fuel Consumption in Mild Alzheimer's Disease
Acronym: MAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-043
Record Dates: First submitted 2016-03-10; First posted 2016-03-15 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2017-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): No intervention
- Physical exercise (Experimental): A 3-month walking program (3 times a week for 12 weeks) on treadmill supervised by a physiotherapist. Duration of the exercise is progressively increased from 15 min to 45 min over a 6-week period and the intensity of the exercise is moderate (a 12-13 score on Borg scale).
  Interventions: Other: Physical exercise

INTERVENTIONS:
Other: Physical exercise — A 3-month walking program (3 times a week for 12 weeks) on treadmill supervised by a physiotherapist. Duration of the exercise is progressively increased from 15 min to 45 min over a 6-week period and the intensity of the exercise is moderate (a 12-13 score on Borg scale).
  Arms: Physical exercise

SUMMARY:
The aim of this study is to evaluate the effect of a 3-month walking program on brain energy metabolism in patient with mild Alzheimer's disease (AD). Two groups of sedentary patients with mild AD are followed and compared over a 3-month period of time: Control (non-active) and walking (from 15 to 45 minutes of exercise on a treadmill, 3 times a week for 12 weeks) groups. All the participants are evaluated on their cognition, brain volumes (MRI) and brain fuel consumption (PET scan with 18-FDG and 11C-AcAc) at the beginning and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild Alzheimer's disease (NINCDS-ADRDA criteria)
* Taking cholinesterase inhibitors
* Sedentary
* Ability to do physical exercise

Exclusion Criteria:

* Parkinson disease
* Down syndrome
* Epilepsy or concussion
* Drug or alcohol abuse
* Past psychiatric history
* Vitamin B12 Deficiency
* Uncontrolled diabetes or thyroid function

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-04; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Paquet, MD, Principal Investigator — Estrie University Integrated Health and Social Services Center - University Hospital of Sherbrooke; Stephen Cunnane, PhD, Principal Investigator — CDRV - CSSS-IUGS - CIUSSS de l'Estrie - CHUS
Locations (1):
- Research Centre on Aging (CSSS-IUGS - CIUSSS de l'Estrie - CHUS), Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Physical Exercise
Started | 3 | 12
Completed | 0 | 10
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Control: The Sedentary group received no active treatment.
- Total: Total of all reporting groups
Arm/Group | Control | Physical Exercise | Total
Number analyzed (Participants) | 3 | 10 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 77 (2) | 73 (4) | 75 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 0 | 4 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Mini-Mental State Examination [Mean (Full Range); unit: points] — The Mini-Mental State Examination (MMSE) is a 30-point questionnaire to measure cognitive impairment. A total score ≥26/30 indicates a normal cognition. Scores below this can indicate mild (20-25 points) , moderate (10-20 points) or severe (≤9 points) cognitive impairment.
  points | 26 [23 to 27] | 26 [23 to 29] | 26 [23 to 29]

OUTCOME MEASURES:

1. Primary Outcome: Brain Glucose Consumption
Description: Brain glucose uptake (umol/100g/min) using 18F-FDG PET imaging
Time Frame: 3 months
Population: Participants of the Control group discontinued the study because of the intense imaging protocol without the possibility of some level of benefit (N=3)
Measure: Mean (Standard Deviation); unit: umol/100 g/min
Arm/Group | Control | Physical Exercise
Number analyzed (Participants) | 0 | 10
umol/100 g/min
  Baseline |  | 27.9 (3.2)
  3-month |  | 28.1 (3.4)

2. Primary Outcome: Brain Acetoacetate Consumption
Description: Brain acetoacetate uptake (umol/100g/min) using 11C-AcAc PET imaging
Time Frame: 3 months
Population: Participants of the Control group discontinued the study because of the intense imaging protocol without the possibility of some level of benefit (N=3). Two participants in the Walking group decided to withdraw from the study prior to the commencement of the exercise program. There were no dropouts over the training period (N=10).
Measure: Mean (Standard Deviation); unit: umol/100 g/min
Arm/Group | Control | Physical Exercise
Number analyzed (Participants) | 0 | 10
umol/100 g/min
  Baseline |  | 0.24 (0.12)
  3-month |  | 0.64 (0.40)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Control Group | Physical Exercise
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-29): https://cdn.clinicaltrials.gov/large-docs/85/NCT02708485/Prot_SAP_000.pdf